CLINICAL TRIAL: NCT06496061
Title: The Efficacy of Adding Leg Wrapping to Prophylactic Norepinephrine Infusion in Reducing the Incidence of Post-spinal Hypotension in Elective Cesarean Section: A PROSPECTIVE DOUBLE- BLINDED RANDOMIZED CLINICAL TRIAL
Brief Title: Leg Wrapping and Norepinephrine for Prevention of Post Spinal Hypotension in C.S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor of Anesthesiology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M728
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Post Spinal Hypotension
Keywords: Post spinal hypotension; Leg wrapping; Prophylactic norepinephrine infusion; Cesarean section
MeSH Terms: interventions — Norepinephrine; Stockings, Compression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leg wrapping and norepinephrine infusion (Experimental): Leg wrapping and norepinephrine infusion. using a crepe bandage (CB) to wrap both legs of the patient from the ankle up to mid-thigh. This CB will be applied tightly enough that the patient feels the tightness but is still comfortable with intact capillary pulsation in the toes and applying norepinephrine infusion 0.5 mg norepinephrine added to 50 ml Normal Saline and set it to run with 0.05 mg/kg/min.
  Interventions: Drug: Norepinephrine; Procedure: Leg wrapping
- Norepinephrine infusion (Active Comparator): Norepinephrine infusion . applying norepinephrine infusion 0.5 mg norepinephrine added to 50 ml Normal Saline and set it to run with 0.05 mg/kg/min.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine infusion with 0.05 mg/kg/h
  Other Names: Noradrenaline infusion
Procedure: Leg wrapping — Elastic leg wrapping
  Other Names: Elastic stockings
  Arms: Leg wrapping and norepinephrine infusion

SUMMARY:
Maternal hypotension after subarachnoid block is considered one of the most common complications that occurs during cesarean delivery, with an incidence of up to 70-80%. Maternal hypotension has adverse effects on both the mother and the fetus such as maternal nausea, vomiting, dizziness, cardiovascular collapse, fetal acidosis, and low Apgar scores).Hence, the prevention of spinal anesthesia-induced hypotension became a topic of great interest for clinicians as well as in literature aiming to improve maternal and neonatal safety. The main etiologies of spinal anesthesia-induced hypotension are aortocaval compression caused by a gravid uterus before delivery of the baby, blood pooling in the lower limbs, and loss of vascular tone as a result of sympatholysis during spinal anesthesia. Based on those mechanisms, Various prophylactic methods have been suggested and tried, including intravenous fluid loading, vasopressors, and physical interventions such as left lateral tilt, leg elevation, and wrapping with crepe bandage (CB). Fluid co-loading with Crystalloids is considered superior to crystalloid preloading and equivalent to colloid preloading. Despite that fluid loading decreased the incidence of hypotension, more interest was directed to vasopressors such as ephedrine, phenylephrine, and norepinephrine. Different regimens have been investigated including continuous infusion or boluses of those vasopressors with promising results reaching lower incidences of hypotension after intrathecal anesthesia but those incidences are still considerable and efforts are made to reach the optimum doses and least hypotension incidences.

Lower limb wrapping with crepe bandages is a simple, non-invasive, nonpharmacological, cost-effective tool that stops blood from pooling in the lower limbs and escaping the central circulation. This method was found to decrease intrathecal-induced hypotension in cesarean delivery to incidences down to 10% in some studies.

We hypothesize that the combination of a pharmacological agent as norepinephrine infusion and a nonpharmacological method as leg wrapping with crepe bandages may help in the prevention of spinal-induced hypotension during Cesarean delivery more than using only one of them.

DETAILED DESCRIPTION:
After the local institutional ethics committee approval, all parturients scheduled for elective Cesarean section at Fayoum University Hospital starting from August 2024 will be enrolled in this prospective randomized study until the completion of the sample size. A detailed written consent will be signed by the eligible parturients before recruitment Parturients will be divided into two groups: (1) Norepinephrine Group (N), 0.05 mg/kg/min, and (2) Norepinephrine & Leg Wrapping Group (NW) Randomization will be done using an online random number generator using a 1:1 ratio. Sequentially numbered sealed opaque envelopes will be opened with each case by an anesthesia resident not involved in patient management. Each envelope contains a code for the group to which this case belongs. The anesthesia resident will follow the instructions within each envelope, cover the lower limbs of the mother, and prepare norepinephrine infusion without further involvement in the study. Pregnant women aged more than 18 years old with a single full-term fetus, scheduled for elective cesarean delivery, will be enrolled in the study. parturients with cardiac Co-morbidities, baseline hypotension with Systolic Blood pressure (SBP) less than 100 mmHg, hypertensive disorders of pregnancy, peripartum bleeding (preoperative placenta Previa or placental abruption), and Body mass index of more than 40 kg/m2, will be excluded. Parturients with Failed intrathecal anesthesia or intraoperative bleeding of more than 500 ml of blood will be excluded from the study. All parturients will be preoperatively assessed and investigated by complete blood count, coagulation profile, Liver and kidney functions. Other investigations as serum electrolytes, ECG, Echocardiography, etc. may be ordered if needed upon case-by case assessment. Pulse oximetry, electrocardiography, and a noninvasive blood pressure cuff will be applied after arrival in the operating room. An 18-gauge cannula will be inserted peripherally, with a stopcock three-way for fluid administration and study infusion. Intravenous 20 mg of Famotidine and 1 mg of Granisetron will be given as a premedication. With the Parturient in the left-lateral tilt position, Baseline SBP will be obtained as the mean of -2-min interval- three consecutive readings. According to each envelope's instructions, the resident will use a crepe bandage (CB) to wrap both legs of the patient from the ankle up to mid-thigh. This CB will be applied with legs raised 45° either (1) loosely in group N, or (2) tightly enough that the patient feels the tightness but is still comfortable with intact capillary pulsation in the toes in group NW. Both lower limbs are then covered from midthigh downwards with surgical drapes. The resident will also prepare the study infusion: 0.5 mg norepinephrine added to 50 ml normal saline and set it to run with 0.05 mg/kg/min. Parturients will then receive intrathecal 11 mg heavy bupivacaine (2.2 ml of 0.5% w/v) with 15 µg of fentanyl by 25-G Quincke spinal needle at L3-4 or L4-5 interspace in the sitting position with rapid crystalloid co-load of 15 ml/kg. After the block, parturients will be positioned in the supine position with left lateral tilt. Pinpricks will be used to assess block success if the sensory level is at T4. The prepared infusion will be started at the same time cerebrospinal fluid is obtained by giving 1 ml bolus followed by the previously calculated rate. This infusion will be continued until five minutes after the delivery of the fetus then it will be stopped gradually over 10 minutes with a decrement decrease of 0.01 mg/kg/min every two minutes. Intraoperative hypertension (defined as an increase in SBP by more than 20% of the baseline) will be managed by temporarily stopping the infusion until systolic blood pressure returns to its normal value. Post-spinal hypotension (defined as a decrease in SBP by more than 20% of the baseline reading during the period from intrathecal injection to delivery) will be managed by 9 mg of IV ephedrine. Severe post-spinal hypotension (defined as a decrease in SBP by more than 40% of the baseline reading) will be managed by 15 mg of IV ephedrine. After two minutes another ephedrine bolus will be given if SBP is not corrected. Intraoperative bradycardia (defined as a heart rate less than 55 beats per minute during the period from intrathecal injection to delivery) associated with hypotension will be managed by 9 mg of IV ephedrine with subsequent 0.5 mg of IV Atropine if bradycardia persists while bradycardia not associated with hypotension will be managed by 0.5 mg of IV Atropine and temporary stopping study infusion until bradycardia resolves. Maternal heart rate will be monitored all through the operation while a noninvasive blood pressure reading will be taken every two minutes starting from intrathecal anesthesia until the end of the operation Co-hydration will be continued up to a maximum of 1.5 l. After delivery oxytocin will be given as a bolus of 0.5 IU over 5 seconds followed by 2.5 IU/h. Our primary outcome is the incidence of post-spinal hypotension. Secondary outcomes include the incidence of severe post-spinal hypotension, hemodynamic data including heart rate and systolic blood pressure at baseline reading and the following 15 readings, time to first hypotensive reading, number of hypotensive episodes, the total dose of ephedrine used, the incidence of hypertension, the incidence of post-delivery hypotension (defined as a decrease in SBP by more than 20% of baseline after delivery of the fetus to the end of the surgery), the incidence of tachycardia, incidence of intraoperative nausea and vomiting, Surgical time (between skin incision and delivery of the fetus), umbilical artery blood gases, and Apgar score for the neonate at 5 min after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged more than 18 years old with a single full-term fetus, scheduled for elective cesarean delivery

Exclusion Criteria:

* parturients with cardiac Co-morbidities, baseline hypotension with Systolic Blood pressure (SBP) less than 100 mmHg, hypertensive disorders of pregnancy, peripartum bleeding (preoperative placenta Previa or placental abruption), and Body mass index of more than 40 kg/m2, will be excluded. Parturients with Failed intrathecal anesthesia or intraoperative bleeding of more than 500 ml of blood

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
the incidence of post-spinal hypotension | From spinal anesthesia to delivery up to 60 minutes
  decrease in SBP by more than 20% of the baseline reading during the period from intrathecal injection to delivery

SECONDARY OUTCOMES:
incidence of sever post-spinal hypotension | From spinal anesthesia to delivery up to 60 minutes
  a decrease in SBP by more than 40% of the baseline reading
total dose of ephedrine | From spinal anesthesia to end of surgery up to 60 minutes
  Amount of ephedrine had been used
incidence of hypertension | From spinal anesthesia to delivery up to 60 minutes
  an increase in SBP by more than 20% of the baseline
incidence of post-delivery hypotension | after delivery to the end of the surgery up to 60 minutes
  a decrease in SBP by more than 20% of baseline
incidence of bradycardia | From spinal anesthesia to end of surgery up to 60 minutes
  heart rate less than 55 beats per minute
Incidence of tachycardia | From spinal anesthesia to end of surgery up to 60 minutes
  Heart rate increased by more than 30% of baseline not related to hypotension or ephedrine use
Incidence of nausea and vomiting | From spinal anesthesia to end of surgery up to 60 minutes
  Nausea and vomiting occuring intraoperative
Umbilical Artery blood gases | From delivery up to 5 minutes
  Measuring pH, pco2,po2 , Hco3 and lactate for umbilical artery blood sample
Apgar score | From delivery up to 5 minutes
  Measuring Apgar score for neonate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JE, George RB, Habib AS. Spinal-induced hypotension: Incidence, mechanisms, prophylaxis, and management: Summarizing 20 years of research. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):57-68. doi: 10.1016/j.bpa.2017.01.001. Epub 2017 Jan 8. PMID 28625306
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Sklebar I, Bujas T, Habek D. SPINAL ANAESTHESIA-INDUCED HYPOTENSION IN OBSTETRICS: PREVENTION AND THERAPY. Acta Clin Croat. 2019 Jun;58(Suppl 1):90-95. doi: 10.20471/acc.2019.58.s1.13. PMID 31741565
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852
- [Background] Tawfik MM, Hayes SM, Jacoub FY, Badran BA, Gohar FM, Shabana AM, Abdelkhalek M, Emara MM. Comparison between colloid preload and crystalloid co-load in cesarean section under spinal anesthesia: a randomized controlled trial. Int J Obstet Anesth. 2014 Nov;23(4):317-23. doi: 10.1016/j.ijoa.2014.06.006. Epub 2014 Jun 30. PMID 25281437
- [Background] Oh AY, Hwang JW, Song IA, Kim MH, Ryu JH, Park HP, Jeon YT, Do SH. Influence of the timing of administration of crystalloid on maternal hypotension during spinal anesthesia for cesarean delivery: preload versus coload. BMC Anesthesiol. 2014 May 16;14:36. doi: 10.1186/1471-2253-14-36. eCollection 2014. PMID 24920942
- [Background] Butwick AJ, Columb MO, Carvalho B. Preventing spinal hypotension during Caesarean delivery: what is the latest? Br J Anaesth. 2015 Feb;114(2):183-6. doi: 10.1093/bja/aeu267. Epub 2014 Jul 30. No abstract available. PMID 25080429
- [Background] Biricik E, Unlugenc H. Vasopressors for the Treatment and Prophylaxis of Spinal Induced Hypotension during Caesarean Section. Turk J Anaesthesiol Reanim. 2021 Feb;49(1):3-10. doi: 10.5152/TJAR.2020.70. Epub 2020 May 5. PMID 33718899
- [Background] Hasanin A, Amin S, Refaat S, Habib S, Zayed M, Abdelwahab Y, Elsayad M, Mostafa M, Raafat H, Elshall A, Fatah SAE. Norepinephrine versus phenylephrine infusion for prophylaxis against post-spinal anaesthesia hypotension during elective caesarean delivery: A randomised controlled trial. Anaesth Crit Care Pain Med. 2019 Dec;38(6):601-607. doi: 10.1016/j.accpm.2019.03.005. Epub 2019 Mar 30. PMID 30935897
- [Background] Prajith KR, Mishra G, Ravishankar M, Hemanth Kumar VR. Hemodynamic changes under spinal anesthesia after elastic wrapping or pneumatic compression of lower limbs in elective cesarean section: A randomized control trial. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):244-250. doi: 10.4103/joacp.JOACP_72_18. Epub 2020 Jun 15. PMID 33013042
- [Background] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625